CLINICAL TRIAL: NCT02404272
Title: Evaluation de la Formation Des infirmières à la Stimulation de l'oralité Des Nouveau-nés Dans Une unité de Réanimation néonatale et Néonatologie : Impact Sur Les Connaissances, Les Pratiques et Sur la qualité Des Soins
Brief Title: Effectiveness of an Oral Feeding Educational Nurse Program on Feeding Performance in Preterm Neonates
Acronym: TOP
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D50855
Record Dates: First submitted 2015-03-13; First posted 2015-03-31 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Preterm Neonates and Feeding
Keywords: Neonate; oral feeding disorder; full oral feeding; training; quality of health care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preterm neonates: All preterm neonates of less than 34 weeks' of gestation admitted to the Neonatology and Neonatal Intensive Care unit of an university hospital located in Lyon, France
  Interventions: Other: Educational oral feeding nurse program

INTERVENTIONS:
Other: Educational oral feeding nurse program — A multidisciplinary group composed of childcare assistants, nurse guardians, speech therapist, physiotherapist, psychologist, and pediatricians will develop and implement the educational oral feeding program. They will provide the 2-day theoretical session as well as the three 2-hour practical sessions including reviews of video recording preterm neonates during bottle or breast feedings.
  The program will focus on non-nutritive sucking for all neonates from 24 up to 34 weeks' of gestation, early oral feeding from 29 weeks' of gestation and oral stimulation for all preterm neonates admitted to the unit. Additionally, all preterm neonates presenting feeding difficulties symptoms will be evaluated weekly by a physiotherapist or speech therapist.
  Each program session is composed of 20 nurses or childcare assistants. Six sessions will be organized in total and all nurses and childcare assistants will be trained

SUMMARY:
Poor oral motor development in preterm neonates is common. Feeding problems lead to longer hospital stay and higher hospital cost. Different interventions have shown their efficacy to accelerate transition and move faster to full oral feeding autonomy. Our study aimed to evaluate the impact of a 2-year education nurse program on feeding pattern and hospital stay of preterm neonates.

This is an interrupted time series study placed in Intensive Care and Neonatal unit of an university hospital located in Lyon, France. All preterm neonates are included in the study, from April 2013 to January 2016.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates of less than 34 weeks' of gestation
* Preterm neonates not requiring surgery with endotracheal intubation
* Preterm neonates hospitalized in the Neonatology and Neonatal Intensive Care Unit of an university hospital, Lyon.
* Preterm neonates discharged from hospital during the study period from April 2013 to January 2016

  --- Exclusion Criteria:
* Preterm neonates presenting delivery age above 34 weeks' of gestation
* Preterm neonates whose parents have expressed their opposition to participate to the study

Ages: 24 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm neonates of less than 34 weeks' of gestation requiring no surgery with endotracheal intubation admitted to the Neonatology or Neonatal Intensive Care Unit of an university hospital, Lyon.
Sampling Method: Non-Probability Sample
Enrollment: 729 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Mean age per month of full oral feeding achievement | Monthly for 34 months
  The age (real and corrected) of weaning of naso-gastric tube of preterm neonates taken out of hospitalization during the month will be computed by subtracting the date of weaning from the date of birth.

SECONDARY OUTCOMES:
Percent of preterm neonates presenting with feeding difficulty symptoms | Monthly for 34 months
  Preterm neonates will be considered as presenting with feeding difficulty symptoms if they present :
  * no demonstration of hunger cues and/or,
  * Coughing,choking or vomiting during bottle or breast feeding and/or,
  * Feed intake exceeding 30 minutes and/or,
  * Excitement, discomfort or arching of the back during feedings and/or,
  * Gagging or falling asleep during feedings and/or,
  * Refusal to feed. The monthly rate of neonates presenting feeding difficulty symptoms will correspond to the total number of neonates presenting feeding difficulty symptoms divided by the number of neonates hospitalized during the month.
Mean length of hospital stay per month | Monthly for 34 months
Morbidity and mortality per month | Monthly for 34 months
  The rate of following neonatal pathologies will be studied :
  * Bronchopulmonary dysplasia,
  * Necrotizing enterocolitis,
  * Periventricular leukomalacia,
  * Intra-ventricular haemorrhage,
  * Premature retinopathy,
  * Hypoxic ischaemic encephalopathy.
Nurses and childcare assistants' satisfaction concerning the educational session | 34 months
  The opinion of nurses and childcare assistants will be collected about the program contents, the organization and the results waited on their practices of care. The qualities of teaching will be assessed by a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne PILLET, Study Director — Hôpital Femme-Mère-Enfant des Hospices Civils de Lyon
Locations (1):
- Hôpital Femme-Mère-Enfant des Hospices Civils de Lyon, Bron, Lyon, France

REFERENCES:
- [Derived] Touzet S, Beissel A, Denis A, Pillet F, Gauthier-Moulinier H, Hommey S, Claris O; TOP Study Group. Effectiveness of a nurse educational oral feeding programme on feeding outcomes in neonates: protocol for an interrupted time series design. BMJ Open. 2016 Apr 15;6(4):e010699. doi: 10.1136/bmjopen-2015-010699. PMID 27084282